CLINICAL TRIAL: NCT07196228
Title: Evaluation of Crestal Bone Changes at Subcrestal Bone-level Implants With Narrow or Regular Tie-base: A Randomized Controlled Trial
Brief Title: Crestal Bone Response to Narrow vs. Regular Tie-Base in Subcrestal Implants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Collaborators: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohammed El-Sawy, Dr, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADMNF-00425
Record Dates: First submitted 2025-09-19; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-01

CONDITIONS: Bone Loss
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Narrow tie-base abutment (Experimental): Patients received subcrestal bone-level implants restored with narrow tie-base abutments.
  Interventions: Device: Intervention Name (Arm 1): Narrow tie-base abutment Intervention Name (Arm 2): Regular tie-base abutment
- Regular tie-base abutment (Placebo Comparator): Patients received subcrestal bone-level implants restored with regular tie-base abutments.
  Interventions: Device: Intervention Name (Arm 1): Narrow tie-base abutment Intervention Name (Arm 2): Regular tie-base abutment

INTERVENTIONS:
Device: Intervention Name (Arm 1): Narrow tie-base abutment Intervention Name (Arm 2): Regular tie-base abutment — Arm 1 - Narrow tie-base abutment
  Intervention Name: Narrow tie-base abutment
  Intervention Type: Device
  Intervention Description: Participants received a subcrestal bone-level dental implant restored with a narrow-diameter tie-base abutment.
  Arm 2 - Regular tie-base abutment
  Intervention Name: Regular tie-base abutment
  Intervention Type: Device
  Intervention Description: Participants received a subcrestal bone-level dental implant restored with a regular-diameter tie-base abutment.

SUMMARY:
This 24-month randomized clinical trial evaluates peri-implant marginal bone changes at subcrestal implants restored with narrow versus regular tie-base abutments.

The study investigates whether narrow or regular tie-base abutments influence peri-implant crestal bone remodeling over 24 months.

This trial assesses the effect of abutment diameter (narrow vs. regular tie-base) on marginal bone stability at subcrestal implants after 24 months.

We aimed to determine if abutment diameter impacts peri-implant marginal bone levels by comparing narrow and regular tie-base abutments in a 24-month RCT.

DETAILED DESCRIPTION:
INTRODUCTION The preservation of supracrestal peri- implant soft tissues plays a crucial role in maintaining bone tissue stability.(1) In recent decades, it has been suggested that peri- implant marginal bone loss is influenced by several factors, including the surface characteristics of the implant neck, the implant- abutment, abutment height, platform switching, and abutment dis/reconnection.(2) Limiting these disconnections has been shown to improve the maintenance of the peri- implant marginal bone level.

On the other hand, it has been observed that transmucosal abutments with convex designs can influence bone remodeling, even with platform switching, when compared to straight or concave abutments.(3,4) The hypothesis was that distancing the abutment- prosthesis interface from the implant shoulder and using narrower transmucosal abutments with platform switching could favor the maintenance of the peri- implant marginal bone level by reducing bone remodeling and the apical migration of the "biological width".

Although there is evidence regarding the influence of platform switching or abutment height on the maintenance of the peri- implant marginal bone level, the evidence on the effect of abutment diameter is limited.(5,6) Therefore, the aim of this 24- month randomized clinical trial is to evaluate changes in the peri- implant marginal bone level at implants restored narrow or regular tie-base after 24 months.

ELIGIBILITY:
**Inclusion Criteria

Adults ≥18 years old.

Single missing tooth in a posterior quadrant, bordered by adjacent natural teeth.

Adequate bone volume to place implants 8.5-10 mm in length and 4 mm in diameter without the need for bone or soft tissue grafting.

Presence of a natural tooth or an implant-supported fixed restoration as an antagonist.

Good oral hygiene with a plaque index <25%.

Willing and able to comply with study procedures and follow-up schedule.

Provided written informed consent.

**Exclusion Criteria

Systemic conditions or medications affecting bone metabolism (e.g., bisphosphonates, corticosteroids).

Untreated periodontitis, persistent oral infections, or poor oral hygiene.

Metabolic bone diseases (e.g., osteoporosis, renal insufficiency, immunodeficiency, leukocyte dysfunction).

History of head and neck radiotherapy.

Physical or mental disability preventing adequate oral hygiene or compliance.

Heavy smoking (>10 cigarettes/day).

Alcoholism or drug abuse.

Pregnancy or breastfeeding.

Bruxism or oral mucosal diseases.

Need for bone regeneration procedures before implant placement.

Inability or unwillingness to attend follow-up visits.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Crestal bone level changes around subcrestal implants | 24 months after loading
  Radiographic assessment of peri-implant marginal bone level changes (in millimeters) comparing narrow versus regular tie-base abutments. Measurements are taken from standardized periapical radiographs at the mesial and distal aspects of each implant, using the implant shoulder as reference.

IPD SHARING:
Plan to Share IPD: No
Up on reasonable request from the corresponding author